CLINICAL TRIAL: NCT04954651
Title: Assessment of the Immunization Levels Against Sars-Cov2 Virus in Subjects Who Have Received European Union (EU) -Approved COVID-19 Vaccines
Brief Title: Assessment of the Immunization Levels Against Sars-Cov2 Virus in Subjects Who Have Received EU-approved COVID-19 Vaccines
Status: Completed | Type: Observational
Sponsor: University of Patras (Other)
Responsible Party: Principal Investigator, Ioannis Habeos, Professor, University of Patras
Other Study IDs: 99-25/2/2021
Record Dates: First submitted 2021-07-06; First posted 2021-07-08 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-06

CONDITIONS: SARS-CoV2 Infection; Vaccine Reaction
Keywords: sars-cov2; vaccine; age
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum from patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- VAC: Vaccinated subject against Sars-Cov2
  Interventions: Biological: Approved vaccines against Sars-Cov2

INTERVENTIONS:
Biological: Approved vaccines against Sars-Cov2 — Subjects who voluntarily are vaccinated against Sars-Cov-2 with any of the approved vaccines by EU

SUMMARY:
Patients who voluntarily visit vaccination centers in Greece against COVID-19 are recruited and their immunization levels against Sars-Cov2 are assesed by measurement of the levels of serum antibodies against Sars-cov-2 before vaccination and in time intervals up to 6-9 months post-vaccination (indicatively 0-1-3-6-9 months post-vaccination).

ELIGIBILITY:
Inclusion Criteria:

* Subjects who voluntarily receive COVID-19 vaccination

Exclusion Criteria:

* Patients who do not complete their vaccination
* Patients who do not provide info on their health status

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects who voluntarily receive COVID-19 vaccines
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2021-07-07 (Actual); Primary Completion 2022-03-28 (Actual); Study Completion 2022-03-28 (Actual)

PRIMARY OUTCOMES:
Antibody titer against Sars-Cov2 | 0-9 months

CONTACTS AND LOCATIONS:
Overall Officials: Ioannis Habeos, MD, PhD, Principal Investigator — University of Patras
Locations (1):
- University Hospital of Patras, Pátrai, Greece

IPD SHARING:
Plan to Share IPD: Undecided
We plan to make the coded individual participant data available to other researchers upon reasonable request after the publication of the study in a journal

REFERENCES:
- [Derived] Parthymou A, Habeos EE, Habeos GI, Deligakis A, Livieratos E, Marangos M, Chartoumpekis DV. Factors associated with anti-SARS-CoV-2 antibody titres 3 months post-vaccination with the second dose of BNT162b2 vaccine: a longitudinal observational cohort study in western Greece. BMJ Open. 2022 May 19;12(5):e057084. doi: 10.1136/bmjopen-2021-057084. PMID 35589363